CLINICAL TRIAL: NCT07235449
Title: Investigation of the Effect of Combined Motor Imagery and Activity Observation Therapy on Strengthening the Non-Dominant Hand in Healthy Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ammar Mahmoud Ahmed, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 61351342/020-1391
Record Dates: First submitted 2025-10-02; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Hand
Keywords: Motor imagery; Action observation; Non-dominant hand; Strengthening exercises
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Motor Imager (Experimental): Conservative Treatment + Motor imagery Program
  Interventions: Other: Conservative treatment + Motor imagery program
- Experimental: Motor imager + Action Observation (Experimental): Conservative Treatment + Motor imagery and Action observation Program
  Interventions: Other: Conservative treatment + Motor imagery and action observation program
- Experimental: Conservative (Active Comparator): Conservative Treatment Program
  Interventions: Other: Conservative treatment via strengthening exercises

INTERVENTIONS:
Other: Conservative treatment + Motor imagery program — Participants will perform guided motor imagery of non-dominant hand strengthening exercises (dumbbell wrist flexion and handball squeeze) without video observation, 5 sessions per week for 4 weeks.
  Arms: Experimental: Motor Imager
Other: Conservative treatment + Motor imagery and action observation program — Participants will observe videos of non-dominant hand strengthening exercises (dumbbell wrist flexion and handball squeeze) and simultaneously perform guided motor imagery of the same movements, 5 sessions per week for 4 weeks.
  Arms: Experimental: Motor imager + Action Observation
Other: Conservative treatment via strengthening exercises — Participants will perform only the physical strengthening exercises (dumbbell wrist flexion and handball squeeze) for the non-dominant hand, 5 sessions per week for 4 weeks, without any motor imagery or action observation.
  Arms: Experimental: Conservative

SUMMARY:
Introduction:

Motor Imagery (MI) and Action Observation (AO) are well-established cognitive training techniques that activate neural networks similar to those involved in actual motor execution. MI involves the mental rehearsal of a movement without physically performing it, while AO relies on observing an action performed by others to stimulate motor-related brain areas. Recent studies suggest that when these methods are combined, they may enhance motor learning, cortical plasticity, and strength gains more effectively than when applied alone. The non-dominant hand, often less trained and weaker in performance compared to the dominant hand, provides an ideal model to examine the effects of these interventions. Strengthening the non-dominant upper limb has implications not only for improving functional balance between the limbs in healthy individuals but also for potential clinical applications in rehabilitation.

Aim:

The primary aim of this randomized controlled study is to investigate the combined effect of MI and AO on muscular strength and functional performance of the non-dominant hand in healthy university students. Specifically, the study seeks to compare the outcomes of three groups: (1) AO combined with MI, (2) MI only, and (3) a control group with no intervention. It is hypothesized that participants in the AO+MI group will demonstrate greater improvements in grip strength and functional outcomes compared to the other groups.

Evaluation:

To comprehensively measure the effects of the intervention, several standardized assessment tools will be employed. Motor imagery ability will be evaluated using the Motor Imagery Questionnaire-3 (MIQ-3). Hand dominance will be determined by the Edinburgh Handedness Inventory. Grip strength will be objectively measured using a Hand Grip Dynamometer. The Recognise App will be used to assess laterality recognition and sensorimotor integration, while overall upper limb function will be measured through the Short Musculoskeletal Function Assessment (SMMT). These evaluations will be conducted both before and after the 4-week intervention period to track changes.

Treatment:

The intervention will span four weeks, with participants attending 2-3 sessions per week. Training protocols will include both cognitive and physical components. In the MI group, participants will engage in guided motor imagery sessions focused on visualizing non-dominant hand exercises. The AO+MI group will observe video demonstrations of the same hand movements, followed by simultaneous motor imagery practice, thereby combining visual and cognitive engagement. Physical strengthening exercises will include dumbbell wrist flexion and handball squeeze, targeting key muscles of the non-dominant hand and forearm. The control group will not undergo any intervention during this period. By integrating AO and MI with specific strengthening exercises, the study aims to determine whether this combined approach enhances neural activation and muscular strength more effectively than MI alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* They agreed to participate
* Having no pathology in hearing and vision
* Having no history of upper limb injury or musculoskeletal
* Having no neurologic disorders
* All subjects had no prior experience with motor imagery
* Having a Standardized Mini-Mental State Test (SMMT) score of more than 24 points

Exclusion Criteria:

* A score of the Movement Imagery Questionnaire (MIQ-3) was less than ≥5
* Severe cognitive deficits
* Neurological problems
* Left-handedness that was measured using the Edinburgh Handedness Inventory

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Handedness was measured using the Edinburgh Handedness Inventory | 3 minutes
  Handedness was measured using the Edinburgh Handedness Inventory, a standardized tool that assesses hand preference in 10 everyday activities (e.g., writing, brushing teeth, using scissors). The Laterality Quotient (LQ) is calculated to determine whether a participant is right-handed, left-handed, or ambidextrous. This measure will be used to identify each participant's dominant and non-dominant hand for the study.
Standardized Mini-Mental State Test | 5 minutes
  The Standardized Mini-Mental State Test (SMMT) is a 30-point cognitive screening tool assessing orientation, memory, attention, language, and visuospatial skills. Scores below 24 indicate cognitive impairment, while scores of 24-30 are considered normal. In this study, the SMMT was used to evaluate cognitive status, and only participants scoring 24 or higher were included.

SECONDARY OUTCOMES:
Movement Imagery Questionnaire (MIQ-3) | 10 minutes
  The Movement Imagery Questionnaire-3 (MIQ-3) is a 12-item tool used to assess an individual's ability to imagine movements through kinesthetic, internal visual, and external visual imagery. Participants physically perform and then imagine specific movements, rating the ease of imagery on a 7-point Likert scale. In this study, the MIQ-3 was used to evaluate motor imagery ability.
Grip Strength Using a hand grip Dynamometer | 8 minutes
  Grip strength, an indicator of upper limb strength and functional capacity, will be measured using a hand grip dynamometer. Participants will sit with the elbow at 90° and wrist in neutral, then squeeze the device maximally for 3-5 seconds. The highest value from 2-3 trials will be recorded as the grip strength score.
Recognize lateralization app | 10 minutes
  The Recognise Hand App (Noigroup) is used to assess left-right hand discrimination and implicit motor imagery ability. Participants view images of hands in different orientations and identify them as left or right, with response time and accuracy recorded. In this study, the app was used to evaluate laterality recognition of the non-dominant hand.

CONTACTS AND LOCATIONS:
Locations (1):
- Ammar Mahmoud Ahmed, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tsukazaki I, Uehara K, Morishita T, Ninomiya M, Funase K. Effect of observation combined with motor imagery of a skilled hand-motor task on motor cortical excitability: difference between novice and expert. Neurosci Lett. 2012 Jun 19;518(2):96-100. doi: 10.1016/j.neulet.2012.04.061. Epub 2012 May 2. PMID 22580208
- [Result] Aoyama T, Kaneko F, Kohno Y. Motor imagery combined with action observation training optimized for individual motor skills further improves motor skills close to a plateau. Hum Mov Sci. 2020 Oct;73:102683. doi: 10.1016/j.humov.2020.102683. Epub 2020 Sep 16. PMID 32949991
- [Result] Marshall B, Wright DJ, Holmes PS, Wood G. Combining Action Observation and Motor Imagery Improves Eye-Hand Coordination during Novel Visuomotor Task Performance. J Mot Behav. 2020;52(3):333-341. doi: 10.1080/00222895.2019.1626337. Epub 2019 Jun 11. PMID 31185831